CLINICAL TRIAL: NCT00782522
Title: Effect Study of an Eccentric Training Program and Stretching for Patients With Chronical Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Special Research Fund, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/380
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Chronical Rotator Cuff Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Eccentric training program
  Interventions: Procedure: Eccentric training program
- 2 (Active Comparator): Traditional training program
  Interventions: Procedure: Traditional training program

INTERVENTIONS:
Procedure: Eccentric training program — Eccentric training program
  Arms: 1
Procedure: Traditional training program — Traditional training program
  Arms: 2

SUMMARY:
In the first part of the the study two new outcome measurements (force reproducibility and subacromial space) will be tested for reproducibility. Therefore 30 healthy people will be assessed.

In a second part of the study 60 patients will be randomly allocated to two groups. Group A (n=30) will perform a traditional training program and group B (n=30) will perform an eccentric training program.

Before the onset of the training programs, pain, function, maximal force, range of motion, subacromial space and force reproducibility will be assessed. Both training programs will be accomplished at home. The first six weeks there will be an appointment with the therapist once a week to explain, correct and when necessary, aggravate the exercises. The next six weeks these appointments will be diminished to once every two weeks.

After 6 and after 12 weeks of training the patients will be reassessed for all the parameters.

ELIGIBILITY:
Inclusion Criteria:

* global tendon thinning
* inhomogeneous echo partitioning
* calcifications at the insertion
* symptoms present for at least 3 months: painful resisted isometric abduction, painful palpation of the supraspinatus tendon, impingement tests positive

Exclusion Criteria:

* documented full thickness rotator cuff rupture
* other lesions than CRCT at the moment of the study
* echographic criteria for ruptures (focal thinning, fluid-filled gap,compressibility)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Maximum force, pain and function,range of motion, force reproduction, subacromial space | After 6 and after 12 weeks of training

CONTACTS AND LOCATIONS:
Overall Officials: Ann Cools, PhD, Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be